CLINICAL TRIAL: NCT00972634
Title: The European Palliative Care Research Collaborative - Computerised Symptom Assessment and Classification of Pain, Depression and Physical Function (Cachexia) (EPCRC - CSA)
Brief Title: Computerized Questionnaires in Assessing Symptoms, Pain, Depression, and Physical Function in Patients With Metastatic and/or Advanced Locoregional Cancer
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: CDR0000648077; NUST-EPCRC-CSA; EU-20962
Record Dates: First submitted 2009-09-04; First posted 2009-09-07 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Cachexia; Depression; Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: depression; cachexia; pain; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Cachexia; Depression; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: computer-assisted intervention — symptom assessment
Other: questionnaire administration — Symptom assessment
Procedure: assessment of therapy complications — Symptom assessment
Procedure: quality-of-life assessment — Symptom assessment

SUMMARY:
RATIONALE: A computer-based system for assessing symptoms may be effective for patients with metastatic or advanced cancer.

PURPOSE: This clinical trial is studying how well computerized questionnaires work in assessing symptoms, pain, depression, and physical function in patients with metastatic and/or advanced local/regional cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility of applying a computer-based system for symptom assessment and classification in palliative cancer care in patients with metastatic and/or advanced cancer.
* Examine hypothesized differences across groups related to acceptance of computers (i.e., age, culture, stage of disease, cognitive and physical function, etc.).
* Examine the general user-friendliness of the tool.
* Test and validate the performance of selected domains and items for classification and assessment of pain and cachexia.
* Explore the validity of domains and items for depression.

OUTLINE: This is a multicenter study.

All patients undergo computer-based assessments of general symptoms by the Edmonton Symptom Assessment System (ESAS) and the European Organization for Research and Treatment of Cancer Core Quality of Life (EORTC QLQ C30) questionnaires and assessment of physical function, appetite/weight loss, and depression by the Brief Patient Health Questionnaire 9 (PRIME-MD PHQ9). Patients who score ≥ 1 (on a 0-10 numerical rating score) on the pain screening question with or without occurrence of breakthrough pain (BTP), undergo the Alberta BTP Assessment tool assessing precipitating factors for pain, time to pain relief after intake of medication, and satisfaction with medication. Patients complete questions regarding user-friendliness and feasibility of using the computer at the end of their session.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of incurable cancer, including patients receiving life-prolonging treatment
* Metastatic and/or advanced locoregional disease

PATIENT CHARACTERISTICS:

* Able to provide written informed consent
* Fluent in the language used at the study site

PRIOR CONCURRENT THERAPY:

* No prior inclusion in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients
Sampling Method: Non-Probability Sample
Enrollment: 1051 (Actual)
Dates: Start 2008-10; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of applying a computer based system for symptom assessment and classification in palliative cancer care | Sept 2008-December 2009
Differences across groups related to acceptance of computers (i.e., age, culture, stage of disease, cognitive and physical function, etc.) | Sept 2008-December 2009
General user-friendliness of the tool | Sept 2008-December 2009
Performance of selected domains and items for classification and assessment of pain and cachexia | Sept 2008-December 2009
Validity of domains and items for depression | Sept 2008-December 2009

CONTACTS AND LOCATIONS:
Overall Officials: Stein Kaasa, MD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Norwegian University of Science and Technology, Trondheim, Norway

REFERENCES:
- [Result] Hjermstad MJ, Lie HC, Caraceni A, Currow DC, Fainsinger RL, Gundersen OE, Haugen DF, Heitzer E, Radbruch L, Stone PC, Strasser F, Kaasa S, Loge JH; European Palliative Care Research Collaborative (EPCRC). Computer-based symptom assessment is feasible in patients with advanced cancer: results from an international multicenter study, the EPCRC-CSA. J Pain Symptom Manage. 2012 Nov;44(5):639-54. doi: 10.1016/j.jpainsymman.2011.10.025. Epub 2012 Jul 13. PMID 22795905
- [Derived] Hjermstad MJ, Kaasa S, Caraceni A, Loge JH, Pedersen T, Haugen DF, Aass N; European Palliative Care Research Collaborative (EPCRC). Characteristics of breakthrough cancer pain and its influence on quality of life in an international cohort of patients with cancer. BMJ Support Palliat Care. 2016 Sep;6(3):344-52. doi: 10.1136/bmjspcare-2015-000887. Epub 2016 Jun 24. PMID 27342412